CLINICAL TRIAL: NCT01284894
Title: Diagnostic Yield of Esophageal High Resolution Manometry in Patients With Unexplained Dysphagia
Brief Title: Esophageal High Resolution Manometry and Dysphagia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2010.624/28
Record Dates: First submitted 2011-01-26; First posted 2011-01-27 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Dysphagia
Keywords: Dysphagia; Conventional manometry; High resolution manometry
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional manometry (Other)
  Interventions: Device: Conventional manometry
- High resolution manometry (Experimental)
  Interventions: Device: High resolution manometry

INTERVENTIONS:
Device: Conventional manometry — Conventional esophageal manometry
  Arms: Conventional manometry
Device: High resolution manometry — High resolution esophageal manometry
  Arms: High resolution manometry

SUMMARY:
Two to 15% of subjects present dysphagia. In case of normal eso-gastro-duodenal endoscopy, patients with dysphagia are referred for esophageal motility testing. Esophageal manometry is the gold standard to evaluate esophageal motility in absence of esophageal obstruction. Two different techniques are available: the conventional manometry and the high resolution manometry. The second one may improve the diagnostic yield and the tolerance of examination in patients with dysphagia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female older than 18 years
* Patient with unexplained dysphagia
* Patient without cause of dysphagia on eso-gastro-duodenal endoscopy
* Patient referred for esophageal manometry
* Patient with health insurance
* Informed consent signed

Exclusion Criteria:

* Patient younger than 18 years
* Allergy to one component of manometry catheter
* Drug intake which can modify the esophageal motricity within 12 hours preceding the realization of the manometry
* Patient unable to give his consent or legally incompetent
* Patient non qualified according to the investigator
* Patient refusal or absence of informed consent signed
* Concomitant participation to another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2011-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Percentage of patients correctly diagnosed for esophageal motility disorder | 6 months

SECONDARY OUTCOMES:
Tolerability (pain, nausea, cough, anxiety) and side effects (nasal bleeding, vomiting, inhalation, esophageal perforation, cardiac failure) | 24 hours
Duration of examination and study analysis | day 0
Cost of patient care within the 6 months following the manometry | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sabine ROMAN, Dr, Principal Investigator — Unité d'Exploration Fonctionnelle Digestive - Hôpital Edouard Herriot - 69437 Lyon Cedex 03- France; Stanislas BRULEY DES VARANNES, Principal Investigator — Service d'Hépato-Gastro-Entérologie - CHU Hôtel Dieu - Place A Ricordeau - 44093 Nantes Cedex - France; Franck ZERBIB, Principal Investigator — Service d'Hépato-Gastro-Entérologie - Hôpital Saint-André - 33075 Bordeaux Cedex - France; Guillaume GOURCEROL, Principal Investigator — Service de Physiologie Digestive, Respiratoire, Urinaire et Sportive - CHU de Rouen - 76031 Rouen Cedex - France; Silvana PERRETTA, Principal Investigator — Pole Hépato- Digestif, Service de Chirurgie digestive et endocrinienne - Nouvel Hôpital Civil - 1 place de l'Hôpital - 67091 Strasbourg cedex - France; Franck ROPERT, Principal Investigator — Service d'Hépato-Gastro-Entérologie - CHU Pontchaillou - Rue H. le Guillou - 35033 Rennes cedex - France; François MION, MD, Principal Investigator — Service d'Hépato-Gastro-Entérologie, Hôpital de la Croix-Rousse , 69317 Lyon; Benoit COFFIN, MD, Principal Investigator — Service d'Hépato-Gastroentérologie, Hôpital Louis Mourier, 92700 Colombes
Locations (1):
- Unité d'Exploration Fonctionnelle Digestive - Hopital Edouard Herriot - 69437 LYON Cedex 03, Lyon, Lyon, France

REFERENCES:
- [Result] Roman S, Huot L, Zerbib F, Bruley des Varannes S, Gourcerol G, Coffin B, Ropert A, Roux A, Mion F. High-Resolution Manometry Improves the Diagnosis of Esophageal Motility Disorders in Patients With Dysphagia: A Randomized Multicenter Study. Am J Gastroenterol. 2016 Mar;111(3):372-80. doi: 10.1038/ajg.2016.1. Epub 2016 Feb 2. PMID 26832656